CLINICAL TRIAL: NCT05269953
Title: A Randomised, Double-blind, Placebo-controlled, Trial of Rhythmic 10Hz Median Nerve Stimulation for the Suppression of the Urge-to-tic and Reduction of Tics in Individuals With Tourette Syndrome and Chronic Tic Disorder
Brief Title: Median Nerve Stimulation for Tourette Syndrome and Chronic Tic Disorder
Acronym: NeSTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Neurotherapeutics Ltd (Unknown); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21NS018
Record Dates: First submitted 2022-01-07; First posted 2022-03-08 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Tourette Syndrome; Chronic Tic Disorder
Keywords: Tourette Syndrome; Median nerve stimulation; Chronic Tic Disorder
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated into three groups (ratio: 1:1:1): active stimulation, sham stimulation and waitlist (no stimulation).
  Those in the waitlist group would receive treatment as normal, prior to an open label phase of receiving active stimulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The member of the research team performing allocation will not be involved in the collection or processing of measurement outcomes (questionnaire/ video data). This same researcher will also be responsible for assigning participants to interventions by programming the MNS devices to deliver sham/active stimulation. This member of the research team will be responsible for creating and maintaining a document which links each participants unique ID with the condition they have been assigned to.
  All other members of the research team, participants and legal guardians will be blind to sham/active group allocation. Participants in the waitlist group and their carers will not be blind to the group they have been allocated to. Participants allocated to the waitlist group will not be blind to the stimulation type they will receive (i.e., all participants initially allocated to the waitlist group will go on to receive active rhythmic MNS at the conclusion of their participation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active stimulation (Experimental)
  Interventions: Device: Active stimulation
- Sham stimulation (Sham Comparator)
  Interventions: Device: Sham stimulation
- Waitlist (no stimulation) (No Intervention): Treatment as usual

INTERVENTIONS:
Device: Active stimulation — Participants assigned to the active stimulation arm will receive rhythmic MNS 2 minutes on and 1 minute off for 15 minutes. The strength of the stimulation will be set to 120% the intensity needed to produce a visible contraction within the thenar muscle.
  Arms: Active stimulation
Device: Sham stimulation — Participants assigned to the sham stimulation arm will receive rhythmic MNS 2 minutes on and 1 minute off for 15 minutes. The strength of the stimulation will be set to 50% the intensity needed to produce a visible contraction within the thenar muscle.
  Arms: Sham stimulation

SUMMARY:
Tourette syndrome (TS) and chronic tic disorder (CTD) are neurodevelopmental disorders that impact approximately 1% of 5-18 year olds worldwide. Both TS and CTD are characterised by the presence of tics, which are repetitive, purposeless, movements or vocalisations of short duration which can occur many times throughout a day. Tics can have a significant negative impact on daily functioning and quality of life, hence, many seek out approaches to manage and reduce their tics and the urges people with TS or CTD often feel preceding them. The two main evidence-based approaches to treating tics are behavioural therapies and medication; both of which can be effective, but accessibility and waitlists are often an issue for behavioural therapies and side effects are common with medication use. Consequently, there is an urgent need for the development of alternative, safe and accessible treatments.

This study aims to examine the effects of rhythmic pulses of electrical stimulation delivered to the wrist in treating tics in people with TS and CTD. In recent work, the investigators have shown that this type of electrical stimulation known as median nerve stimulation (MNS), can substantially reduce tics and related urges during stimulation. The investigators now want to extend this work to examine the effects of the stimulation on a higher number of people, compared to placebo and treatment as usual. The investigators will do this through assessment of symptom change using questionnaires, interviews and videos collection during four weeks of stimulation and two time points afterwards.

The investigators have developed a new MNS device for this trial which is portable and easy to use. The primary hypothesis is that active rhythmic MNS will lead to a reduction in tic severity compared to a placebo condition. The secondary hypothesis is that MNS will also have a positive beneficial effect on urges, impairment, well-being and co-occurring Obsessive-Compulsive Disorder (OCD) symptoms compared to both sham stimulation and no stimulation.

DETAILED DESCRIPTION:
The symptoms of Tourette Syndrome (TS) (tics and premonitory urges) can be treated using behavioural therapies and/or medications, however access, availability, side effects and treatment resistance are factors which many people with TS and their family's express frustration with. Therefore, it is in the interest of patients and the wider medical community that alternative treatments are tested and scientifically validated. In recent work, the investigators have found that low intensity electrical stimulation delivered to the wrist can be effective in significantly reducing tics and tic related premonitory urges. In the study the investigators want to expand this work to examine the effects of the stimulation on a higher number of people, compared to placebo and treatment as usual and to examine the suitability of a wearable device for delivering stimulation from home.

The investigators will conduct a parallel, double-blind, placebo-controlled trial of a wearable, wrist-worn, therapeutic device for the suppression of premonitory urge and the reduction of tics in individuals with TS. In order to validate the device as a genuine and effective form of therapy, it is essential that a placebo branch of the study is completed. Participants will be made aware of the three different experimental arms ahead of enrolment and will be debriefed following completion of the trial. The investigators are committed to clearly explaining why a placebo condition is essential, while minimising the amount of information the investigators withhold from participants, hence the investigators feel it is important to be able to let participants know the condition participants were in at the end of the trial.

The device the investigators are aiming to trial will be programmed to deliver low-intensity (1-19 mA) rhythmic (10Hz) trains of electrical stimulation to the median nerve for 14 minutes, and will be used by each participant from home once each day, 5 days each week, for a period of 4 weeks. Participants assigned to the active condition will experience rhythmic (10Hz) trains of stimulation set to an individual intensity which the investigators have found to be effective in the investigators' previous work (-120% of intensity needed to generate a visible muscle twitch in the thenar muscle). Those assigned to the placebo group will receive stimulation at a subthreshold rate (50% intensity needed to generate thenar muscle twitch). The investigators' previous work suggests that this serves as a sufficient control condition. Those in the waitlist group would receive treatment as normal, prior to an open label phase of receiving active stimulation.

A total of 135 participants (45 per group) will be allocated to one of the three groups; active stimulation; sham stimulation; or waitlist (i.e., treatment as usual). In order to minimise the difference in age, gender and symptom severity between groups, the investigators will perform a stratified randomisation for age, gender and severity (using Yale Global Tic Severity Scale (YGTSS) Total Tic Severity Score) to allocate individuals to each group.

The effects of the stimulation will be assessed using several semi-structured interviews, questionnaire measures and video recordings of participant's tics. The investigators will also use questionnaire measures/ interviews to measure baseline characteristics of the participants, as these factors may influence response to the investigators proposed intervention. The majority of this trial will be remotely supervised and therefor the majority of these measures will also be taken through video call and online questionnaire measures with the exception of an initial visit to the University of Nottingham.

The primary hypothesis is that active MNS will lead to a reduction in tic severity compared to subthreshold placebo stimulation. The procedure for testing this will be as follows:

1. Participants who have expressed an interest in the study will be given a detailed participant information sheet. Participants will be given the opportunity to ask questions about the study. If participants wish to proceed and to have an initial telephone screening to assess eligibility participants will then be asked to complete an initial consent form which will asked for their consent to take part in the screening and for the research team to keep a record of their answers during that process.
2. Consenting participants will then be contacted by a member of the research team at an agreed time via telephone/video call. This call should last no longer than an hour. This will be used to give participants further insights into the trial and to establish trial eligibility. Trial eligibility will be assessed according to the investigators' predefined inclusion/ exclusion criteria. The YGTSS, semi structured interview will also be conducted by a trained member of the research team to establish If the potential participant has enough tics to be eligible for the trial.
3. After completing the telephone screening, eligible participants will be sent a further electronic consent form to take part in the rest of the trial. After obtaining consent, participants will be allocated into a trial arm and a date will be set for them to visit Nottingham. In the case of the wait list group participants will not visit Nottingham until participants have entered into the open label active phase of the trial.
4. During the baseline visit to the University of Nottingham, participants will receive the stimulation device and will be trained in its correct placement and use. In order to ensure participant's comfort with the stimulation, a practice session will be performed. If the participant experiences significant discomfort, participants will be withdrawn from the trial. On the same day, demographic information along with primary and secondary measures will be collected using various questionnaires and structured interviews. Participants in the waitlist group will also complete these measurements online and through video call.
5. Participants in the active and placebo groups will return home with the device and be instructed to commence stimulation sessions on the following Monday. Participants will be asked to use the device once each day, 5 days each week, for a period of 4 weeks. During the stimulation period participants will be asked to complete a few short questions each day which should take 1-2 minutes. Participants will also be contacted by a member of the research team at weeks 1, 2, 3 and 4 of stimulation and 3 and 6 months after completing stimulation. During these meetings through video call lasting approximately 1 hour various semi-structured interviews and questionnaires will be administered to assess changes in symptoms. A subset of participants will also be asked to record videos of themselves 5 minutes before the stimulation, during the stimulation and 5minutes after the stimulation and to upload these to a secure online platform. These will be used by the research team to objectively count changes in tics.

The investigators estimate that the trial will take 9 months to collect all data sets, including the 6 month follow up period. Visits to Nottingham will take place during the first 3 months of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 years or older. Must also be able to give informed consent (along with parents/guardians).
* Confirmed or suspected diagnosis of Tourette Syndrome or Chronic Tic Disorder with a moderate amount of tics (to be assessed during an initial screening interview).
* Stable treatment regime/no treatment for the past 2 months (i.e. if taking medication same drug & dosage).
* Internet access & access to electronic device to complete online questionnaires and video calls.
* Participants must be able to travel to Nottingham for one visit and have reliable access to the internet.
* Participant is willing and able to give informed consent for participation in the clinical investigation.
* Able (in the Investigators opinion) and willing to comply with all clinical investigation requirements
* Resident in the UK

Exclusion Criteria:

* Current diagnosis of epilepsy.
* Participant or participants guardian (if under 16) unable to read/write in English.
* Participants will be excluded from the trial if they find the stimulation too uncomfortable during a practice session at the in person baseline visit.
* Individuals with implanted electronic devices (e.g. pacemakers, insulin pump, implantable cardioverter defibrillator, neurostimulators).
* Individuals sharing the household with an individual with implanted electronic devices (e.g. pacemakers, insulin pump, implantable cardioverter defibrillator, neurostimulators).
* Individuals with current/ recent diagnosis or symptoms of SARS-CoV-2 will not be invited to visit the university until it is safe for them to do so (2 weeks following positive test).
* Individuals with a diagnosis of non-verbal autism or similar condition which would affect ability to give informed consent to take part in the study will not be recruited.
* Pregnant women will not be recruited for this study.
* Participants who have participated in previous research studies involving median nerve stimulation
* Participants aged over 90 years old

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Change in Yale Global Tic Severity Scale - revised (YGTSS-R) total tic severity score | Baseline, week 1, 2, 3 and 4, and at follow-up points 3 and 6 months after starting stimulation
  The primary outcome measure will be the scores from our core measures of tic severity (using scores from YGTSS-R). The YGTSS-R total tic severity score range from 0-50, where higher scores indicate a worse outcome. These will be used to assess any change in tic severity symptoms between groups and over the initial 4 week stimulation period.

SECONDARY OUTCOMES:
Change in Premonitory urge for Tics Scale-Revised (PUTS-R) | Baseline, week 1, 2, 3 and 4, and at follow-up points 3 and 6 months after starting stimulation
  This outcome measure will evaluate treatment effects of MNS on the occurrence of the urge-to-tic by looking at change in scores from the PUTS. The PUTS scores range from 0-32, where higher scores indicate a worse outcome.
Change in Tic impairment (as measured through subscales of YGTSS-R) | Baseline, week 1, 2, 3 and 4, and at follow-up points 3 and 6 months after starting stimulation
  This outcome measure will evaluate the treatment effects of MNS on tic related impairment by looking at change in scores from the Tic impairment subscale in the YGTSS-R. Tic impairment score range from 0-50, where higher scores indicate a worse outcome.
Change in Quality of life (as measured by Gilles de la Tourette Syndrome - Quality of Life scale (GTS-QoL)) | Baseline, week 4, and at follow-up points 3 and 6 months after starting stimulation
  This outcome measure will evaluate the treatment effects of MNS on well-being by looking at change in scores from the GTS-QoL. The GTS-QoL scores range from 0-100, where higher scores indicate worse outcome. This questionnaire includes a visual analog scale ranging 0-100 assessing how satisfied the person feels in their life, higher scores indicating a better outcome.
Change in Anxiety symptoms (as measured by Becks anxiety inventory (BAI)) | Baseline, week 4, and at follow-up points 3 and 6 months after starting stimulation
  This outcome measure will evaluate the treatment effects of MNS on co-occurring Anxiety symptoms by looking at change in scores from the BAI. The BAI scores range from 0-63, where higher scores indicate worse outcome.
Change in OCD symptoms as measured by (Children's) Yale-Brown Obsessive-Compulsive Scale ((C)Y-BOCS) | Baseline, week 1, 2, 3 and 4, and at follow-up points 3 and 6 months after starting stimulation
  This outcome measure will evaluate the treatment effects of MNS on co-occurring OCD symptoms by looking at changes in scores from the (C)Y-BOCS. The (C)Y-BOCS scores range from 0-40, where higher scores indicate worse outcome.
Change in Tic frequency as quantified by analysis of video data | Daily during the first 2 weeks of stimulation
  This outcome measure will explore the changes in tic frequency occurring during and immediately following MNS, through the use of video data in a subgroup of participants

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Colin Campbell Building, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeon S, Walkup JT, Woods DW, Peterson A, Piacentini J, Wilhelm S, Katsovich L, McGuire JF, Dziura J, Scahill L. Detecting a clinically meaningful change in tic severity in Tourette syndrome: a comparison of three methods. Contemp Clin Trials. 2013 Nov;36(2):414-20. doi: 10.1016/j.cct.2013.08.012. Epub 2013 Aug 31. PMID 24001701
- [Background] Robertson MM, Eapen V, Cavanna AE. The international prevalence, epidemiology, and clinical phenomenology of Tourette syndrome: a cross-cultural perspective. J Psychosom Res. 2009 Dec;67(6):475-83. doi: 10.1016/j.jpsychores.2009.07.010. PMID 19913651
- [Background] Cohen SC, Leckman JF, Bloch MH. Clinical assessment of Tourette syndrome and tic disorders. Neurosci Biobehav Rev. 2013 Jul;37(6):997-1007. doi: 10.1016/j.neubiorev.2012.11.013. Epub 2012 Dec 1. PMID 23206664
- [Background] Cavanna AE, Black KJ, Hallett M, Voon V. Neurobiology of the Premonitory Urge in Tourette's Syndrome: Pathophysiology and Treatment Implications. J Neuropsychiatry Clin Neurosci. 2017 Spring;29(2):95-104. doi: 10.1176/appi.neuropsych.16070141. Epub 2017 Jan 25. PMID 28121259
- [Background] Leckman JF, Walker DE, Cohen DJ. Premonitory urges in Tourette's syndrome. Am J Psychiatry. 1993 Jan;150(1):98-102. doi: 10.1176/ajp.150.1.98. PMID 8417589
- [Background] Freeman RD, Fast DK, Burd L, Kerbeshian J, Robertson MM, Sandor P. An international perspective on Tourette syndrome: selected findings from 3,500 individuals in 22 countries. Dev Med Child Neurol. 2000 Jul;42(7):436-47. doi: 10.1017/s0012162200000839. PMID 10972415
- [Background] Conelea CA, Woods DW, Zinner SH, Budman C, Murphy T, Scahill LD, Compton SN, Walkup J. Exploring the impact of chronic tic disorders on youth: results from the Tourette Syndrome Impact Survey. Child Psychiatry Hum Dev. 2011 Apr;42(2):219-42. doi: 10.1007/s10578-010-0211-4. PMID 21046225
- [Background] Conelea CA, Woods DW, Zinner SH, Budman CL, Murphy TK, Scahill LD, Compton SN, Walkup JT. The impact of Tourette Syndrome in adults: results from the Tourette Syndrome impact survey. Community Ment Health J. 2013 Feb;49(1):110-20. doi: 10.1007/s10597-011-9465-y. Epub 2011 Nov 4. PMID 22052430
- [Background] Robertson MM. Mood disorders and Gilles de la Tourette's syndrome: An update on prevalence, etiology, comorbidity, clinical associations, and implications. J Psychosom Res. 2006 Sep;61(3):349-58. doi: 10.1016/j.jpsychores.2006.07.019. PMID 16938513
- [Background] Fernandez de la Cruz L, Rydell M, Runeson B, Brander G, Ruck C, D'Onofrio BM, Larsson H, Lichtenstein P, Mataix-Cols D. Suicide in Tourette's and Chronic Tic Disorders. Biol Psychiatry. 2017 Jul 15;82(2):111-118. doi: 10.1016/j.biopsych.2016.08.023. Epub 2016 Aug 26. PMID 27773353
- [Background] Whittington C, Pennant M, Kendall T, Glazebrook C, Trayner P, Groom M, Hedderly T, Heyman I, Jackson G, Jackson S, Murphy T, Rickards H, Robertson M, Stern J, Hollis C. Practitioner Review: Treatments for Tourette syndrome in children and young people - a systematic review. J Child Psychol Psychiatry. 2016 Sep;57(9):988-1004. doi: 10.1111/jcpp.12556. Epub 2016 May 2. PMID 27132945
- [Background] Roessner V, Plessen KJ, Rothenberger A, Ludolph AG, Rizzo R, Skov L, Strand G, Stern JS, Termine C, Hoekstra PJ; ESSTS Guidelines Group. European clinical guidelines for Tourette syndrome and other tic disorders. Part II: pharmacological treatment. Eur Child Adolesc Psychiatry. 2011 Apr;20(4):173-96. doi: 10.1007/s00787-011-0163-7. PMID 21445724
- [Background] Hollis C, Pennant M, Cuenca J, Glazebrook C, Kendall T, Whittington C, Stockton S, Larsson L, Bunton P, Dobson S, Groom M, Hedderly T, Heyman I, Jackson GM, Jackson S, Murphy T, Rickards H, Robertson M, Stern J. Clinical effectiveness and patient perspectives of different treatment strategies for tics in children and adolescents with Tourette syndrome: a systematic review and qualitative analysis. Health Technol Assess. 2016 Jan;20(4):1-450, vii-viii. doi: 10.3310/hta20040. PMID 26786936
- [Background] Azrin NH, Nunn RG. Habit-reversal: a method of eliminating nervous habits and tics. Behav Res Ther. 1973 Nov;11(4):619-28. doi: 10.1016/0005-7967(73)90119-8. No abstract available. PMID 4777653
- [Background] Piacentini J, Woods DW, Scahill L, Wilhelm S, Peterson AL, Chang S, Ginsburg GS, Deckersbach T, Dziura J, Levi-Pearl S, Walkup JT. Behavior therapy for children with Tourette disorder: a randomized controlled trial. JAMA. 2010 May 19;303(19):1929-37. doi: 10.1001/jama.2010.607. PMID 20483969
- [Background] Cuenca J, Glazebrook C, Kendall T, Hedderly T, Heyman I, Jackson G, Murphy T, Rickards H, Robertson M, Stern J, Trayner P, Hollis C. Perceptions of treatment for tics among young people with Tourette syndrome and their parents: a mixed methods study. BMC Psychiatry. 2015 Mar 11;15:46. doi: 10.1186/s12888-015-0430-0. PMID 25879205
- [Background] Hsu CW, Wang LJ, Lin PY. Efficacy of repetitive transcranial magnetic stimulation for Tourette syndrome: A systematic review and meta-analysis. Brain Stimul. 2018 Sep-Oct;11(5):1110-1118. doi: 10.1016/j.brs.2018.06.002. Epub 2018 Jun 5. PMID 29885862
- [Background] Charvet LE, Shaw MT, Bikson M, Woods AJ, Knotkova H. Supervised transcranial direct current stimulation (tDCS) at home: A guide for clinical research and practice. Brain Stimul. 2020 May-Jun;13(3):686-693. doi: 10.1016/j.brs.2020.02.011. Epub 2020 Feb 10. PMID 32289698
- [Background] Fregni F, El-Hagrassy MM, Pacheco-Barrios K, Carvalho S, Leite J, Simis M, Brunelin J, Nakamura-Palacios EM, Marangolo P, Venkatasubramanian G, San-Juan D, Caumo W, Bikson M, Brunoni AR; Neuromodulation Center Working Group. Evidence-Based Guidelines and Secondary Meta-Analysis for the Use of Transcranial Direct Current Stimulation in Neurological and Psychiatric Disorders. Int J Neuropsychopharmacol. 2021 Apr 21;24(4):256-313. doi: 10.1093/ijnp/pyaa051. PMID 32710772
- [Background] Morera Maiquez B, Sigurdsson HP, Dyke K, Clarke E, McGrath P, Pasche M, Rajendran A, Jackson GM, Jackson SR. Entraining Movement-Related Brain Oscillations to Suppress Tics in Tourette Syndrome. Curr Biol. 2020 Jun 22;30(12):2334-2342.e3. doi: 10.1016/j.cub.2020.04.044. Epub 2020 Jun 4. PMID 32502412
- [Background] Houlgreave MS, Morera Maiquez B, Brookes MJ, Jackson SR. The oscillatory effects of rhythmic median nerve stimulation. Neuroimage. 2022 May 1;251:118990. doi: 10.1016/j.neuroimage.2022.118990. Epub 2022 Feb 11. PMID 35158022
- [Background] Armstrong S, Sale MV, Cunnington R. Neural Oscillations and the Initiation of Voluntary Movement. Front Psychol. 2018 Dec 18;9:2509. doi: 10.3389/fpsyg.2018.02509. eCollection 2018. PMID 30618939
- [Background] Debes N, Jeppesen S, Raghava JM, Groth C, Rostrup E, Skov L. Longitudinal Magnetic Resonance Imaging (MRI) Analysis of the Developmental Changes of Tourette Syndrome Reveal Reduced Diffusion in the Cortico-Striato-Thalamo-Cortical Pathways. J Child Neurol. 2015 Sep;30(10):1315-26. doi: 10.1177/0883073814560629. Epub 2014 Dec 22. PMID 25535056